CLINICAL TRIAL: NCT07175597
Title: Trial of Acceptability, Tolerability and Biochemical Indicators of Hibiscus Sabdariffa L. Drink in Pregnant Women
Brief Title: Pilot Trial of Hibiscus Drink During Pregnancy (PTHDDP)
Acronym: PTHDDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Victor Eduardo Alcantar Rodríguez (Other)
Collaborators: National Polytechnic Institute, Mexico (Other)
Responsible Party: Sponsor-Investigator, Victor Eduardo Alcantar Rodríguez, Associate Research Professor B, National Polytechnic Institute, Mexico
Organization: National Polytechnic Institute, Mexico (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IPNMexico
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pregnant Woman
Keywords: Functional foods; Hibiscus sabdariffa drink; Pilot 1 clinical trial; Hypertension; Biomarkers
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Four-week phase I pilot trial where participants are their own controls with pre- and post-treatment measurements
Masking Description: This trial included only one group, assessing the acceptability and tolerability of a beverage, as well as its effects on markers. The results will be used to promote a study with a larger number of participants and a longer timeframe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Experimental): Pregnant women in the second trimester of pregnancy who consumed a daily dose of Hibiscus sabdariffa drink for 4 weeks
  Interventions: Dietary Supplement: Hibiscus sabdariffa drink

INTERVENTIONS:
Dietary Supplement: Hibiscus sabdariffa drink — A daily dose of Hibiscus sabdariffa drink that provides 9.6 mg of anthocyanins

SUMMARY:
The goal of this phase I pilot clinical trial is to evaluate the acceptability, tolerability and effect on blood pressure and biomarkers of Hibiscus sabdariffa drink in pregnant women in the second trimester of pregnancy. The main questions it aims to answer are:

Is the drink acceptable to take as a daily dose for a long time? Does drinking the beverage cause negative effects? What is the effect of drink consumption on blood pressure and biomarkers in pregnant women?

Each participant was their own control with the values measured before consumption of the beverage and after four weeks of consumption.

The participants:

* Took a daily dose of the beverage for 4 weeks
* Once a week for the four weeks, they answered the acceptability and tolerability questionnaires
* Before starting to consume the beverage and after the 4 weeks of consumption, they had their blood pressure measured, and samples taken for biomarker measurements.

ELIGIBILITY:
Inclusion Criteria:

* Women in the second trimester of pregnancy (14 to 28 gestation weeks)
* Age 18 to 35 years
* Blood pressure <140/90 mmHg

Exclusion Criteria:

* Multiple or high-risk pregnancy
* Hypertensive disorder in previous pregnancies
* Body mass index >32 kg/m2
* Present chronic diseases

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of Hibiscus sabdariffa drink | 4 weeks
  Beverage acceptability was measured using a sensory evaluation with 7-point hedonic scale of the attributes of odor, color, flavor, mouthfeel, aftertaste, and overall appearance through questionnaires applied once a week for 4 weeks.
  The outcome measures are based on a 7-point hedonic scale where every participant can answer in every attribute evaluated:
  1. I dislike it a lot
  2. I dislike it moderately
  3. I dislike it a little
  4. I neither like it nor dislike it
  5. I like it a little
  6. I like it moderately
  7. I like it a lot
Tolerability of Hibiscus sabdariffa Drink | 4 weeks
  Tolerability was measured by the presence or absence of gastrointestinal symptoms such as nausea, regurgitation, vomiting, constipation, diarrhea, flatulence, and abdominal pain through questionnaires applied once a week for 4 weeks.
  The outcome measures for the tolerability assessment were the presence or absence of gastrointestinal symptoms mentioned in the previous paragraph, where participants had the option to respond:
  1. Symptom absent
  2. Symptom present but not bothersome
  3. Symptom present and somewhat bothersome, but does not interfere with daily activities or sleep
  4. Symptom present and bothersome because it interferes with daily activities or sleep
  5. Required medical attention

SECONDARY OUTCOMES:
Blood pressure | 4 weeks
  Blood pressure was measured using the Korotkoff auscultation method, These measurements were taken before starting to consume the beverage and at the end of the 4-week trial.
  The outcome measures were the average of the measurements of the 10 participants expressed as mm/Hg of systolic and diastolic pressure.
Biomarkers glucose | 4 weeks
  Glucose was measured by taking a blood sample, These measurements were taken before starting to consume the beverage and at the end of the 4-week trial.
  The outcome measures were the average of the measurements of the 10 participants expressed as mg/dL.
Biomarkers cholesterol | 4 weeks
  Cholesterol was measured by taking a blood sample, These measurements were taken before starting to consume the beverage and at the end of the 4-week trial.
  The outcome measures were the average of the measurements of the 10 participants expressed as mg/dL.
Biomarkers triglycerides | 4 weeks
  Triglycerides were measured by taking a blood sample, These measurements were taken before starting to consume the beverage and at the end of the 4-week trial.
  The outcome measures were the average of the measurements of the 10 participants expressed as mg/dL.
Biomarkers creatinine | 4 weeks
  Creatinine was measured by taking a blood sample, These measurements were taken before starting to consume the beverage and at the end of the 4-week trial.
  The outcome measures were the average of the measurements of the 10 participants expressed as mg/dL.
Biomarkers proteinuria | 4 weeks
  Participants were also asked to provide a urine sample to determine proteinuria.
  These measurements were taken before starting to consume the beverage and at the end of the 4-week trial.
  The results were presented as the number of positive cases for proteinuria, as well as the average of positive cases expressed as mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Victor E. Alcantar Rodríguez, PhD Student, Principal Investigator — National Polytechnic Institute and Autonomous University of Barcelona
Locations (1):
- MEDOMAI, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: Yes
A platform will be sought to publish the results databases.
Supporting Information: Study Protocol, ICF, CSR

DOCUMENTS (2):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT07175597/Prot_000.pdf
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT07175597/ICF_001.pdf